CLINICAL TRIAL: NCT04949178
Title: Impact of Continuous Renal Replacement Therapy on Systemic Hemodynamics and Lactate Clearance in Critically Ill Cirrhotics With Septic Shock.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-41
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood and urine sample (~10 ml) would be stored for assessing the serum cytokine profile, endotoxin levels, NT-Pro BNP, Troponin I levels, urine N-GAL before, 6 hours and at 24 hours after initiation of CRRT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill cirrhotics with septic shock and AKI undergoing CRRT: Consecutive critically ill cirrhotics with septic shock and AKI who give written informed consent will be included in this prospective study
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study.

SUMMARY:
Consecutive critically ill cirrhotics with septic shock and AKI who give written informed consent will be included in this prospective study. A blood and urine sample (~10 ml) would be stored for assessing the serum cytokine profile, endotoxin levels, NT-Pro BNP, Troponin I levels, urine N-GAL before, 6 hours and at 24 hours after initiation of CRRT. Septic shock will be defined by the presence of two or more diagnostic criteria for the systemic inflammatory response syndrome, proven or suspected infection with hypotension non-responsive to adequate fluid resuscitation assessed by no evidence of stroke volume variation on flow track and need of a vasopressor to achieve a target mean arterial pressure (MAP) of ≥ 65 mm Hg. A record of SVR, SVRI, global ejection fraction, extravascular lung water index and pulmonary vascular permeability index, CVP, IVC diameter and B-lines on ultrasound lung would be recorded. A record of the clearance of lactate at 6, 12 , 24 and daily till recovery or death would be performed. Patients with age less than 18 years, severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD) pregnancy, chronic kidney disease on hemodialysis, extremely moribund patients with an expected life expectancy of less than 24 hours, failure to give informed consent from family members.

DETAILED DESCRIPTION:
AIM: Assessment of the impact of CRRT on systemic hemodynamics and microcirculation in critically ill cirrhotics with septic shock and AKI.

Primary Objective To study the impact of continuous renal replacement therapy on systemic hemodynamics (improvement in systemic vascular resistive index, cardiac index) and lactate clearance in critically ill cirrhotics with septic shock.

Secondary Objectives Impact on endothelial function and inflammatory cytokines Impact on renal functions and ammonia Incidence of hemodynamic instability and/or intradialytic hypotension Impact on lung injury scores (as determined by EVLW and PVPI) To study the duration of mechanical ventilation and ICU stay Impact on transplant-free survival To evaluate the improvement in SOFA, MELD and APACHE scores.

Methodology: Consecutive critically ill cirrhotics with septic shock and AKI who give written informed consent will be included in this prospective study. A blood and urine sample (~10 ml) would be stored for assessing the serum cytokine profile, endotoxin levels, NT-Pro BNP, Troponin I levels, urine N-GAL before, 6 hours and at 24 hours after initiation of CRRT. Septic shock will be defined by the presence of two or more diagnostic criteria for the systemic inflammatory response syndrome, proven or suspected infection with hypotension non-responsive to adequate fluid resuscitation assessed by no evidence of stroke volume variation on flow track and need of a vasopressor to achieve a target mean arterial pressure (MAP) of ≥ 65 mm Hg. A record of SVR, SVRI, global ejection fraction, extravascular lung water index and pulmonary vascular permeability index, CVP, IVC diameter and B-lines on ultrasound lung would be recorded. A record of the clearance of lactate at 6, 12 , 24 and daily till recovery or death would be performed. Patients with age less than 18 years, severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD) pregnancy, chronic kidney disease on hemodialysis, extremely moribund patients with an expected life expectancy of less than 24 hours, failure to give informed consent from family members.

Study Design:

Prospective observational cohort study

Study Population: Critically ill cirrhotics with septic shock and AKI undergoing CRRT

Study Period: May 2021- December 2021

Sample size: It will be time based study with a minimum sample size of 50 patients. Currently, there is no study looking at these outcomes in critically ill cirrhotics.

Intervention: (Not a part of the study protocol), Patients on Continuous Renal Replacement Therapy (CRRT) will be enrolled.

Monitoring and Assessment: Hourly till the time patient is on dialysis then as indicated.

Adverse Effects: Worsening of hypotension, sepsis, bleeding, allergic reactions to dailyser, any cardiac side-effects.

Statistical analysis

* All variables shall be expressed in mean (sd) or median (range)
* Variables will be compared by Mann- Whitney U test
* For Categorical variables we will use Chi-Square or Fisher's test
* Survival analysis will be done using cox-proportional regression analysis

Actuarial probability of survival shall be calculated by Kaplan- Meier graph and compared by log- rank test.

Stopping rule: Unstable hemodynamics, worsening of shock and lactic acidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Critically ill cirrhotics undergoing continuous renal replacement therapy.

Exclusion Criteria:

1. Patients with age less than 18 years
2. Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
3. Pregnancy
4. Chronic kidney disease on hemodialysis
5. Extremely moribund patients with an expected life expectancy of less than 24 hours
6. Failure to give informed consent from family members.
7. Hemodynamic instability requiring very high dose of vasopressors.
8. Septic shock would be defined as clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP>=65 mm of Hg and having a serum lactate >2 mmol/L despite adequate volume resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill cirrhotics with septic shock and AKI undergoing CRRT
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-25 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of SVR from baseline by 20% or above 600 and decrease in vasopressors at 24 hours after CRRT initiation. | 24 hours

SECONDARY OUTCOMES:
Lactate clearance after CRRT initiation | 6 hours
Lactate clearance after CRRT initiation | 12 hours
Lactate clearance after CRRT initiation | 24 hours
Incidence of renal recovery | 24 hours
Incidence of dialysis associated complications (hypotension, bleeding, hypothermia, catheter-related blood stream infections would be recorded). | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India